CLINICAL TRIAL: NCT05727176
Title: Phase 2 Study of Futibatinib 20 mg and 16 mg in Patients With Advanced Cholangiocarcinoma With FGFR2 Fusions or Rearrangements
Brief Title: Study of Futibatinib in Patients With Advanced Cholangiocarcinoma With FGFR2 Fusion or Rearrangement
Acronym: FOENIX-CCA4
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-205; 2023-503665-39 (EudraCT Number); 2022-9400 (Other: Japan PMDA CTN Receipt Number)
Expanded Access: NCT04507503 (Approved for marketing)
Record Dates: First submitted 2023-01-23; First posted 2023-02-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cholangiocarcinoma; FGFR2 Fusions; Gene Rearrangement
Keywords: Futibatinib; Advanced cholangiocarcinoma; cholangiocarcinoma; FGFR2; Fusion; Rearrangemen; TAS-120
MeSH Terms: conditions — Cholangiocarcinoma | interventions — futibatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): TAS-120 (20mg) tablets, oral; 21-day cycle
  Interventions: Drug: TAS-120
- Treatment Arm B (Experimental): TAS-120 (16mg) tablets, oral; 21-day cycle
  Interventions: Drug: TAS-120

INTERVENTIONS:
Drug: TAS-120 — TAS-120 is an oral FGFR inhibitor
  Other Names: Futibatinib

SUMMARY:
This is an open-label, multinational, randomized Phase 2 study confirming the clinical benefit of 20 mg futibatinib and evaluating the safety and efficacy of 16 mg futibatinib in previously treated CCA harboring FGFR2 gene fusions and other rearrangements.

DETAILED DESCRIPTION:
This is an open-label, multinational, randomized Phase 2 study confirming the clinical benefit of 20 mg futibatinib and evaluating the safety and efficacy of 16 mg futibatinib in previously treated CCA harboring FGFR2 gene fusions and other rearrangements. Eligible patients will be randomized on a 1:1 basis to the following study arms:

* Patients will receive futibatinib at an oral dose of 16 mg, administered daily (QD) on every day of a 21-day cycle.
* Patients will receive futibatinib at an oral dose of 20 mg, administered daily (QD) on every day of a 21-day cycle.

Patients may continue to receive continuous futibatinib until documentation of progressive disease (PD) per RECIST 1.1, or until other withdrawal criteria are met, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, locally advanced, metastatic, or unresectable intrahepatic of extrahepatic Cholangiocarcinoma.
2. Documented evidence of FGFR2 gene fusions or other FGFR2 rearrangement
3. Received at least one prior systemic gemcitabine and platinum-based regimen for CCA
4. Documentation of radiographic disease progression on the most recent prior therapy
5. Measurable disease
6. performance status 0 or 1
7. Adequate organ function

Exclusion Criteria:

1. History or current evidence of calcium and phosphate homeostasis disorder
2. Current evidence of clinically significant retinal disorder
3. Treatment with any of the following within the specified time frame prior to the first dose of futibatinib:

   1. Major surgery within the previous 4 weeks (the surgical incision should be fully healed prior to the first dose of futibatinib) and radiotherapy for extended field within 4 weeks or limited field radiotherapy within 2 weeks
   2. Patients with locoregional therapy, eg, transarterial chemoembolization (TACE), selective internal radiotherapy (SIRT) or ablation within 4 weeks
   3. Any non investigational anticancer therapy within 3 weeks or have not recovered from side effects of such therapy prior to futibatinib. Endocrine therapy is allowed for patients with breast or prostate cancer
   4. Targeted therapy or immunotherapy within 3 weeks or within 5 half lives Any investigational agent received within 5 half-lives of the drug or 4 weeks, whichever is shorter.
   5. Patients with prior FGFR-directed therapy
4. A serious illness or medical condition(s) including (but not limited to) the following:

   1. Known brain metastasis (not including primary brain tumors) unless patient is clinically stable for ≥1 month
   2. Known acute systemic infection
   3. Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV New York Heart Association [NYHA] Classification) within the previous 2 months; if >2 months, cardiac function must be within normal limits and the patient must be free of cardiac-related symptoms
   4. Significant gastrointestinal disorder(s) that could interfere with the absorption of futibatinib.
   5. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the Investigator would make the patient inappropriate for entry into this study.
5. Known additional malignancy that is progressing or requires active treatment, with the exception of patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or antitumor assessment of the investigational regimen. Exceptions must be discussed with the Sponsor prior to patient enrollment.
6. Pregnant or lactating female.
7. Known hypersensitivity or severe reaction to futibatinib or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR by independent central review | 12 months after the study completion
  defined as the proportion of patients experiencing a best overall response of partial response (PR) or complete response (CR) (per RECIST 1.1), based on ICR

SECONDARY OUTCOMES:
DoR by independent review | up to 12 months after the study completion
  defined as time from the first documentation of response to the first documentation of objective tumor progression by ICR (per RECIST 1.1) or death due to any cause, whichever occurs first
PFS by independent review | up to 12 months after the study completion
  defined as the time from date of randomization to the date of documentation of disease progression by ICR per RECIST (version 1.1, 2009) or date of death, whichever comes first
ORR per Investigator assessment | up to 12 months after the study completion
  defined as proportion of patients experiencing a best overall response of partial response (PR) or complete response (CR) (per RECIST v1.1).
DoR per Investigator assessment | up to 12 months after the study completion
  defined as time from the first documentation of response to the first documentation of objective tumor progression or death due to any cause, whichever occurs first
PFS per Investigator assessment | up to 12 months after the study completion
  defined as the time from date of randomization to the date of disease progression based on Investigator assessment of radiographic images or death, whichever occurs first
OS | up to 12 months after the study completion
  defined as the time from the date of randomization until the date of death due to any cause.
Treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0 | up to 12 months after the study completion
  Safety will be assessed based on reported AEs (including SAEs), graded by CTCAE V5.0. including serious adverse events (SAEs) and dose modifications.
Change from Baseline in Quality of life as assessed by EORTC QLQ-C30 | up to 12 months after the study completion
  Change from Baseline in quality of life as assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score
Change from Baseline in Quality of life as assessed by EuroQol-5D (EQ-5D ) | up to 12 months after the study completion
  Change from Baseline in Quality of Life as Assessed by European Quality of Life - 5 Dimensions-3 Levels (EQ-5D-3L) Scale Score.

CONTACTS AND LOCATIONS:
Locations (65):
- United States (10):
  - University of California San Diego UCSD - Moores Cancer Center, La Jolla, California
  - Tampa General Hospital Cancer Institute, Tampa, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Gabrail Cancer Center Research, Canton, Ohio
  - Texas Oncology, Abilene, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Texas Oncology Methodist DFW, Dallas, Texas
  - Texas Onc Methodist (Charlton), Dallas, Texas
  - Texas Oncology - Northeast, Denton, Texas
  - Center for Oncology and Blood Disorders, Houston, Texas
- Argentina (3):
  - Hospital Britanico, Buenos Aires
  - CEMIC, CABA
  - Sanatorio de la Mujer, Rosario
- Australia (3):
  - St Vincent's Hospital Sydney - The Kinghorn Cancer Centre, Sydney, New South Wales
  - Alfred Health, Medical Oncology Unit, Second floor William Buckland Radiotherapy Center, Melbourne, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Brazil (5):
  - Instituto do Cancer do Estado de Sao Paulo, Cerqueira César
  - IOP - Instituto de Oncologia do Parana, Curitiba
  - Hospital Erasto Gaertner, Curitiba
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
  - Fundacao Antonio Prudente - A.C.Camargo Cancer Center, São Paulo
- Canada (4):
  - Grand River Hospital - Grand River Regional Cancer Centre (GRRCC), Kitchener, OH
  - Sunnybrook Health Sciences Center, Toronto, OH
  - University of Toronto, Toronto, OH
  - McGill University Health Center, Montreal, Quebec
- China (10):
  - Guangdong Provincial People's Hospitall, Guangzhou, Guangdong
  - Harbin Medical University - Cancer Hospital, Harbin, Heilongjiang
  - Jiangsu Provance Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong University - Shandong Cancer Hospital, Jinan, Shandong
  - Zhongahan Hospital Fudan unversity, Shanghai, Shanghai Municipality
  - West China Hospital- Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Shanghai Gobroad Cancer Hospital China Pharmaceutical University, Shanghai
  - Tongji University Shanghai East Hospital, Shanghai
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong Island
  - The Chinese University of Hong Kong Prince of Wales Hospital, New Territories
- Italy (3):
  - Policlinico S. Orsola-Malpighi, Bologna
  - IRCCS Humanitas Research Hospital, Rozzano
  - AOUI Verona - Ospedale Borgo Roma, Verona
- Japan (5):
  - Tohoku University Hospital, Sendai, Miyagi
  - National Cancer Center Hospital East, Kashiwa-Shi
  - Nagasaki University Hospital, Nagasaki
  - Nagoya University Hospital, Nagoya
  - Osaka Metropolitan University Hospital, Osaka-Fu
- Poland (4):
  - Szpital Wojewdzki w Koszalinie im. Mikoaja Kopernika, Koszalin
  - Centrum Onkologii Ziemi Lubelskiej im. w. Jana z Dukli, Lublin
  - Europejskie Centrum Zdrowia Otwock Sp. Z.o.o., Otwock
  - Centrum Onkologii-Instytut im. Marii Skłodowskiej - Curie, Warsaw
- Portugal (2):
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar Lisboa Norte CHLN EPE - Hospital de Santa Maria, Lisbon
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, Seongnam
  - Yonsei University Health System - Severance Hospital, Seoul
  - The Catholic University of Korea, St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia de l'Hospitalet de Llobregat - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra, Medical Oncology Service (Mariano Ponz Sarvise), Madrid
  - Hospital Universitario Fundación Jimenez Díaz, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No